CLINICAL TRIAL: NCT04394377
Title: Randomized Clinical Trial to Evaluate a Routine Full Anticoagulation Strategy in Patients With Coronavirus (COVID-19) - COALIZAO ACTION Trial
Brief Title: Full Anticoagulation Versus Prophylaxis in COVID-19: COALIZAO ACTION Trial
Acronym: ACTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital do Coracao (Other); Hospital Sirio-Libanes (Other); Hospital Moinhos de Vento (Other); Hospital Alemão Oswaldo Cruz (Other); Beneficência Portuguesa de São Paulo (Other); Brazilian Research In Intensive Care Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002/2020
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Infection
Keywords: SARS-CoV2; Anticoagulation; Coronavirus infection; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): The routine full anticoagulation strategy will be applied for 30 days. In this strategy, full anticoagulation therapy will be maintained for all patients randomized to group 1 and, depending on the patient's clinical condition, there will be 2 possible routes of administration (oral or parenteral):
  * Oral: Rivaroxaban 20 mg 1 x daily (adjust the dose to 15 mg 1x daily if ClCr between 30 and 49ml/min and/or concomitant use of azithromycin);
  * Parenteral: Enoxaparin 1 mg/kg every 12 hours subcutaneously or Unfractionated heparin (preferable option for patients progressing with disseminated intravascular coagulation).
  Interventions: Drug: Group 1: Rivaroxaban 20mg/d followed by enoxaparin/unfractionated heparin when needed
- Group 2 (Other): Patients in this group will receive the usual standard management and currently have no indication of full anticoagulation. Venous thromboembolism (VTE) prophylaxis should be used in group 2 (usual standard of care) as recommended by guidelines.
  Interventions: Drug: Group 2: control group with enoxaparin 40mg/d

INTERVENTIONS:
Drug: Group 1: Rivaroxaban 20mg/d followed by enoxaparin/unfractionated heparin when needed — Routine full anticoagulation strategy
  Arms: Group 1
Drug: Group 2: control group with enoxaparin 40mg/d — Usual standard of care and currently have no indication of full anticoagulation.
  Arms: Group 2

SUMMARY:
Pragmatic randomized clinical trial of patients admitted to the hospital with confirmed COVID-19 infection and elevated D-Dimer.

Randomization 1:1 - Group 1 will undergo a routine full anticoagulation (oral or parenteral when needed) strategy; and group 2 will receive usual standard of care with prophylactic anticoagulation

DETAILED DESCRIPTION:
Patients admitted to hospital with confirmed COVID-19, and who meet the eligibility criteria will be invited to participate in the proposed study. Following the application of the informed consent form, they will collect the D-dimer (if they have not yet collected it routinely from the hospital) and confirm the value over the normal limit in patients with confirmed COVID-19, will be randomized to 2 groups in the 1:1 ratio. Group 1 will follow the strategy of routine use of full anticoagulation therapy (oral or parenteral when indicated); and group 2 will follow the usual standard care with in-hospital prophylactic anticoagulation (without routine full anticoagulation).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of COVID-19 admitted to hospital;
* Duration of symptoms related to hospitalization ≤ 14 days;
* Patients ≥ 18 year old;
* D-dimer above the upper limit of normal (collected until 72 hours before the randomization);
* Agreement to participate by providing the informed consent form (ICF).

Exclusion Criteria:

* Patients with indication for full anticoagulation during inclusion (for example, diagnosis of venous thromboembolism, atrial fibrillation, mechanical valve prosthesis);
* Platelets < 50,000 /mm3
* Need for ASA therapy > 100 mg;
* Need for P2Y12 inhibitor therapy (clopidogrel, ticagrelor or prasugrel);
* Chronic use of non-hormonal anti-inflammatory drugs;
* Sustained uncontrolled systolic blood pressure (BP) of ≥180 mmHg or diastolic BP of ≥100 mmHg;
* INR > 1,5;
* Patients contraindicated to full anticoagulation (active bleeding, liver failure, blood dyscrasia or prohibitive hemorrhage risk as evaluated by the investigator);
* Criteria for disseminated intravascular coagulation (DIC);
* A history of hemorrhagic stroke or any intracranial bleeding at any time in the past or current intracranial neoplasm (benign or malignant), cerebral metastases, arteriovenous (AV) malformation, or aneurysm;
* Active cancer (excluding non-melanoma skin cancer) defined as cancer not in remission or requiring active chemotherapy or adjunctive therapies such as immunotherapy or radiotherapy;
* Hypersensitivity to rivaroxaban;
* Use of strong inhibitors of cytochrome P450 (CYP) 3A4 and/or P-glycoprotein (P-gp) (e.g. protease inhibitors, ketoconazole, Itraconazole) and/or use of P-gp and strong CYP3A4 inducers (such as but not limited to rifampin/rifampicin, rifabutin, rifapentine, phenytoin, phenobarbital, carbamazepine, or St. John's Wort);
* Known HIV infection;
* Creatinine clearance < 30 ml/min according to the Cockcroft-Gault Formula;
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Hierarchical composite endpoint composed of mortality, number of days alive, number of days in the hospital and number of days with oxygen therapy at the end of 30 days. | In 30 days
  The primary objective will be analyzed using the win ratio approach comparing every participant of treatment group to every participant of control group to determine a winner.

SECONDARY OUTCOMES:
Incidence of Venous thromboembolism | In 30 days
Incidence of acute myocardial infarction | In 30 days
Incidence of stroke | In 30 days
Number of days using oxygen therapy | In 30 days
Peak of troponin | In 30 days
Peak of D-dimer | In 30 days
Incidence of Major bleeding and clinically relevant non-major bleeding by the ISTH criteria | In 30 days
  It will be considered the main safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Renato D. Lopes, MD, PhD, Study Chair — BCRI
Locations (36):
- Brazil (36):
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Centro de Ensino e Aperfeiçoamento em Pesquisa - CEAP, Serra, Espírito Santo
  - Centro de Estudos Clínicos do Hospital Cárdio Pulmonar, Salvador, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Santa Casa de Misericórdia da Bahia - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Centro de Pesquisas Cardiológicas de Goiânia do Hospital das Clínicas (UFG), Goiânia, Goiás
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Núcleo de Ciências de Saúde - Unidade de Pesquisa - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Clínica do Hospital de Clínicas da Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Hospital Universitário da Universidade Estadual de Londrina, Londrina, Paraná
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Instituto Baia Sul de Ensino E Pesquisa Dr. Irineu May Brodbeck / Hospital Baía Sul, Florianópolis, Santa Catarina
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Hospital de Amor de Barretos - (Pio XII), Barretos, São Paulo
  - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - Unesp, Botucatu, São Paulo
  - Hospital Universitário São Francisco de Assis, Bragança Paulista, São Paulo
  - Hospital Regional do Litoral Norte, Caraguatatuba, São Paulo
  - Hospital Regional de Registro, Registro, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - Centro Integrado de Pesquisa (CIP) - Hospital de Base de Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Regional de São José dos Campos, São José dos Campos, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga, São Paulo
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - Hcor - Hospital do Coração, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Moriah, São Paulo
  - Hospital Samaritano Paulista, São Paulo
  - Hospital Santa Paula, São Paulo
  - Hospital São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual de S. Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP-InCor-HCFMUSP, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All data provided during study is anonymized to respect the privacy of patients who have participated in the trial in line with applicable regulations.

REFERENCES:
- [Derived] de Barros E Silva PGM, Furtado RHM, de Alcantara Chaud MS, Macedo AVS, Bronhara B, Damiani LP, Barbosa LM, Suiama MA, Ramacciotti E, de Aquino Martins P, de Oliveira AL, Nunes VS, Ritt LEF, Rocha AT, Tramujas L, Santos SV, Diaz DRA, Viana LS, Melro LMG, Figueiredo EL, Neuenschwander FC, Dracoulakis MDA, Lima RGSD, de Souza Dantas VC, Fernandes ACS, Gebara OCE, Hernandes ME, Queiroz DAR, Veiga VC, Canesin MF, de Faria LM, Feitosa-Filho GS, Gazzana MB, Liporace IL, de Oliveira Twardowsky A, Maia LN, Machado FR, de Matos Soeiro A, Conceicao-Souza GE, Armaganijan L, Guimaraes PO, Rosa RG, Azevedo LCP, Alexander JH, Avezum A, Berwanger O, Cavalcanti AB, Lopes RD; ACTION Coalition COVID-19 Brazil IV Investigators. Predictors of bleeding and thrombotic events among patients admitted to the hospital with COVID-19 and elevated D-dimer: insights from the ACTION randomized clinical trial. J Thromb Thrombolysis. 2024 Aug;57(6):1031-1039. doi: 10.1007/s11239-024-02995-y. Epub 2024 May 18. PMID 38762708
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Lopes RD, de Barros E Silva PGM, Furtado RHM, Macedo AVS, Bronhara B, Damiani LP, Barbosa LM, de Aveiro Morata J, Ramacciotti E, de Aquino Martins P, de Oliveira AL, Nunes VS, Ritt LEF, Rocha AT, Tramujas L, Santos SV, Diaz DRA, Viana LS, Melro LMG, de Alcantara Chaud MS, Figueiredo EL, Neuenschwander FC, Dracoulakis MDA, Lima RGSD, de Souza Dantas VC, Fernandes ACS, Gebara OCE, Hernandes ME, Queiroz DAR, Veiga VC, Canesin MF, de Faria LM, Feitosa-Filho GS, Gazzana MB, Liporace IL, de Oliveira Twardowsky A, Maia LN, Machado FR, de Matos Soeiro A, Conceicao-Souza GE, Armaganijan L, Guimaraes PO, Rosa RG, Azevedo LCP, Alexander JH, Avezum A, Cavalcanti AB, Berwanger O; ACTION Coalition COVID-19 Brazil IV Investigators. Therapeutic versus prophylactic anticoagulation for patients admitted to hospital with COVID-19 and elevated D-dimer concentration (ACTION): an open-label, multicentre, randomised, controlled trial. Lancet. 2021 Jun 12;397(10291):2253-2263. doi: 10.1016/S0140-6736(21)01203-4. Epub 2021 Jun 4. PMID 34097856
- [Derived] Lopes RD, de Barros E Silva PGM, Furtado RHM, Macedo AVS, Ramacciotti E, Damini LP, Bronhara B, Cavalcanti AB, Rosa RG, Azevedo LCP, Veiga VC, Machado FR, Ritt LE, Martins PA, Alexander JH, Avezum A, Berwanger O; Coalition COVID-19 Brazil IV Investigators. Randomized clinical trial to evaluate a routine full anticoagulation Strategy in Patients with Coronavirus Infection (SARS-CoV2) admitted to hospital: Rationale and design of the ACTION (AntiCoagulaTlon cOroNavirus)-Coalition IV trial. Am Heart J. 2021 Aug;238:1-11. doi: 10.1016/j.ahj.2021.04.005. Epub 2021 Apr 20. PMID 33891907
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773